CLINICAL TRIAL: NCT05975346
Title: Evaluation of the Efficacy of Preoperative Ketamine Nebulization on Postoperative Sore Throat Due to Tracheal Intubation for Adult Patients Under General Anesthesia, A Prospective Randomized Controlled Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Doaa Ahmed Abdellatif, Resident-anesthesia,ICU and pain manegment department-sohag hospital university, Sohag University
Other Study IDs: soh-Med-23-07-20MS
Record Dates: First submitted 2023-07-27; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Post Operative Sore Throat
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- (K) Ketamine group: 40 patients will receive ketamine 50mg (1.0 ml with 4.0 ml of the saline) nebulization
  Interventions: Drug: Ketamine
- (S) Saline group: 40 patients will receive saline nebulization (5ml).
  Interventions: Other: saline nebulization

INTERVENTIONS:
Drug: Ketamine — description
  Groups: (K) Ketamine group
Other: saline nebulization — description
  Groups: (S) Saline group

SUMMARY:
Sore throat includes specific symptoms such as dysphagia, dysphonia, hoarseness, continuous throat pain, and pharyngeal dryness. Patients rated postoperative sore throat (POST) as the eighth most undesirable outcome in the postoperative period POST has a reported incidence of up to 62% following general anesthesia (GA). The incidence of POST is more common in GA with tracheal intubation than in GA with the supraglottic airway Ketamine is an N-methyl-D-aspartate (NMDA) receptor antagonist and has been used as a gargle for reducing the incidence and severity of POST due to its anti-nociceptive and anti-inflammatory effects

ELIGIBILITY:
Inclusion Criteria:

1. Age 16-60 years.
2. Of both sex.
3. American Society of Anesthesiologists Physical Status (ASA PS) I-II.
4. Undergoing general anesthesia with endotracheal intubation with surgery duration less than two hours.

Exclusion Criteria:

* a- History of chronic obstructive History of sore throat or upper respiratory tract infection.

  b- Intraoral and intrapharyngeal surgery. c- airway disease or Asthma. d- Mallampati grade more than II. e- Known allergic to study drug. f- More than one attempt is required for intubation. g- Hypertensive patients. h- Epileptic patients. i- cerebral palsy or any neurological disorders. j- Psychiatry patients. k- Cardiac patients. l- Perioperative use of anti-inflammatory drugs (Non-steroidal anti-inflammatory drug or steroids).

Ages: 16 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: 1. Age 16-60 years.
  2. Of both sex.
  3. American Society of Anesthesiologists Physical Status (ASA PS) I-II.
  4. Undergoing general anesthesia with endotracheal intubation with surgery duration less than two hours.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
the incidence and severity of POST | at immediate recovery (0 h), 2, 4, 6, 8, 12 and 24 h post-operatively.
  the study is to measure the incidence and severity of POST at immediate recovery (0 h), 2, 4, 6, 8, 12 and 24 h post-operatively. in adult patients undergoing surgery of a duration less than 2h.

SECONDARY OUTCOMES:
evaluation of side effects including nausea, vomiting, cough, and dry mouth in both groups. | at immediate recovery (0 h), 2, 4, 6, 8, 12 and 24 h post-operatively.
  evaluation of side effects including nausea, vomiting, cough, and dry mouth in both groups.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cairns A, Battleday FM, Velikova G, Brunelli A, Bell H, Favo J, Patella M, Lindner O, Pompili C. General patient satisfaction after elective and acute thoracic surgery is associated with postoperative complications. J Thorac Dis. 2020 May;12(5):2088-2095. doi: 10.21037/jtd-19-3345b. PMID 32642112
- [Background] Hailu S, Shiferaw A, Regasa T, Getahun YA, Mossie A, Besha A. Incidence of Postoperative Sore Throat and Associated Factors Among Pediatric Patients Undergoing Surgery Under General Anesthesia at Hawassa University Comprehensive Specialized Hospital, a Prospective Cohort Study. Int J Gen Med. 2023 Feb 18;16:589-598. doi: 10.2147/IJGM.S397519. eCollection 2023. PMID 36845340
- [Background] Thomas D, Bejoy R, Zabrin N, Beevi S. Preoperative ketamine nebulization attenuates the incidence and severity of postoperative sore throat: A randomized controlled clinical trial. Saudi J Anaesth. 2018 Jul-Sep;12(3):440-445. doi: 10.4103/sja.SJA_47_18. PMID 30100844